CLINICAL TRIAL: NCT00928330
Title: A Phase Ib, Open-Label Study of the Safety, Tolerability, Pharmacokinetics, and Activity of Trastuzumab and Trastuzumab-MCC-DM1 Administered Intravenously and GDC-0941 Administered Orally to Patients With HER2-Positive Metastatic Breast Cancer Who Have Progressed on Previous Trastuzumab-Based Therapy
Brief Title: Trastuzumab and Trastuzumab-MCC-DM1 Administered Intravenously and GDC-0941 Administered Orally to Patients With HER2-Positive Metastatic Breast Cancer Who Have Progressed on Previous Trastuzumab-Based Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDC4627g; GO01302 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Metastatic Breast Cancer
Keywords: TDM-1; HER2; HER2+; HER2+ Breast Cancer; HER-2; MBC; Trastuzumab emtansine
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Trastuzumab; Ado-Trastuzumab Emtansine

ARMS (3):
- A (Experimental)
  Interventions: Drug: GDC-0941; Drug: trastuzumab-MCC-DM1
- B (Experimental)
  Interventions: Drug: GDC-0941; Drug: trastuzumab-MCC-DM1
- C (Experimental)
  Interventions: Drug: GDC-0941; Drug: Trastuzumab

INTERVENTIONS:
Drug: GDC-0941 — Oral repeating dose
Drug: Trastuzumab — Intravenous repeating dose
  Arms: C
Drug: trastuzumab-MCC-DM1 — Intravenous repeating dose
  Arms: A; B

SUMMARY:
This multicenter, Phase Ib study is an open label, dose escalation, three-arm study evaluating the safety, tolerability, pharmacokinetics, and activity of oral (PO) GDC 0941 administered in combination with either intravenous (IV) infusion of T-DM1 or IV infusion of trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally advanced or metastatic breast cancer that has progressed on at least one trastuzumab-based regimen in the metastatic or locally advanced setting
* HER2-positive disease documented by one of the following results using FDA-approved testing methods: FISH-positive, chromogenic in situ hybridization (CISH)-positive, or IHC 3 + by local laboratory assessment
* Life expectancy >= 90 days
* Agreement to use an effective form of contraception for the duration of the study

Exclusion Criteria:

* History of Grade >= 3 hypersensitivity reaction to trastuzumab, or Grade >= 1 with the most recent trastuzumab infusion before study entry, or continued requirement for prolonged trastuzumab infusions to prevent hypersensitivity reactions
* History of intolerance to trastuzumab and/or adverse events related to trastuzumab that resulted in trastuzumab being permanently discontinued
* Prior anti-cancer therapy (e.g., biologic or other targeted therapy, chemotherapy, hormonal therapy) within 2 weeks prior to Day 1
* Prior investigational anti-cancer therapy within 4 weeks prior to Day 1
* Grade >= 2 peripheral neuropathy
* History of Grade >= 3 hyperglycemia (fasting)
* History of Type 1 or Type 2 diabetes requiring daily medication
* History of clinically significant cardiac or pulmonary dysfunction
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with HIV, hepatitis B virus, or hepatitis C virus
* Any condition requiring anticoagulants, such as warfarin, heparin, or thrombolytic agents
* Any condition requiring > 2 grams of acetaminophen daily
* Need for current chronic corticosteroid therapy
* Pregnancy, lactation, or breast-feeding
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1, or anticipation of the need for major surgery during the course of study treatment
* Symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac function | Through study completion or early study discontinuation
Changes in vital signs, physical findings, and clinical laboratory results during and following administration of study drugs that result in dose modification, dose delay, or discontinuation of T-DM1 and/or GDC 0941 | Through study completion or early study discontinuation
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
PK parameters of T-DM1 and GDC-0941 (total exposure, maximum serum concentration, and minimum concentration) | Through study completion or early study discontinuation
Progression-free survival (PFS) | From study treatment initiation to the first occurrence of disease progression or death on study
Objective response based on investigator assessment | Confirmed response >/= 4 weeks after initial documentation of response
Duration of response | Time from initial complete or partial response to the time of disease progression or death on study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (3):
- United States (3):
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts